CLINICAL TRIAL: NCT04335929
Title: Internet-based Cognitive Behavioural Therapy for Spanish Tinnitus Sufferers: A Global Pilot Trial
Brief Title: Internet-based Cognitive Behavioural Therapy for Spanish Tinnitus Sufferers
Acronym: ICBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lamar University (Other)
Responsible Party: Principal Investigator, Vinaya Manchaiah, Jo Mayo Endowed Professor, Lamar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY20-200-2
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based Cognitive Behavior Therapy (Experimental): The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.
  Interventions: Behavioral: Internet-based Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavior Therapy — The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.

SUMMARY:
Nearly 50 million people in the U.S. experience tinnitus, of which about 20 million people have burdensome chronic tinnitus. Tinnitus can be very debilitating as many aspects of daily life can be affected, such as sleep, mood, and concentration. Currently, there is no cure for tinnitus. Pharmacological or sound-therapy based interventions are sometimes provided but may be of limited value to certain individuals. Research suggests that Cognitive Behavior Therapy (CBT) based approaches have the most evidence of effectiveness in the management of tinnitus. However, CBT is rarely offered to tinnitus sufferers in the U.S. (less than 1%), partly because of lack of trained professionals who can deliver CBT. To improve access to CBT for tinnitus, an online CBT program has been developed which is also available in Spanish. However, the outcomes of the Spanish version of the program has not been evaluated. The purpose of the current study is to determine the feasibility of guided Spanish version of the Internet-based CBT (ICBT) using audiological support on tinnitus distress and tinnitus-related comorbidities.

DETAILED DESCRIPTION:
Objective: The purpose of the current study is to determine the feasibility of guided Spanish version of the Internet-based CBT (ICBT) using audiological support on tinnitus distress and tinnitus-related comorbidities.

Hypothesis: It is hypothesized that Spanish version of the ICBT will reduce the tinnitus-related distress, decrease sleep disturbance, decrease anxiety and depression, and improve health-related quality of life in Spanish speaking tinnitus suffers. The investigators also hypothesize that these results will be stable in both short- and long-term post-intervention.

Design: A single group assignment, with a one-year follow-up design will be used to evaluate the feasibility of Spanish version of the ICBT on tinnitus distress.

Setting: This will be an Internet-based study for Spanish speaking tinnitus suffers living across the globe.

Participants: Eligible participants will include adults with tinnitus for a minimum period of 3 months with internet access and no major medical or psychiatric conditions. 50 Spanish speaking participants will be recruited.

Intervention: The intervention offered is a guided CTB-based internet intervention (ICBT), providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.

Outcome measures: The main outcome measure is the Tinnitus Functional Index (TFI). Secondary outcome measures are the Tinnitus and Hearing Survey (THS), Tinnitus Cognition Questionnaire (TCQ), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), Insomnia Severity Index (ISI), and EuroQol EQ-5D-5L VAS.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years and older adults from across the globe;
2. the ability to read and type in Spanish;
3. no barriers to using a computer (e.g. no significant fine motor control or visual problems);
4. Internet and e-mail access and the ability to use it;
5. commitment to completing the program;
6. completion of the online screening and outcome questionnaires;
7. agree to participate in either group and be randomized to one of these groups;
8. understand and work towards the end goal of reducing the impact and distress of tinnitus, although the strength of the tinnitus may remain the same;
9. be available for 12 months after starting the study to complete a 1-year follow-up questionnaire; and
10. experience bothersome tinnitus for a minimum period of 3 months;

Exclusion Criteria:

1. reporting any major medical or psychiatric conditions;
2. reporting pulsatile, objective or unilateral tinnitus, which has not been investigated medically;
3. tinnitus as a consequence of a medical disorder, still under investigation; and
4. undergoing any other tinnitus therapy while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Manchaiah, PhD, Principal Investigator — Lamar University
Locations (1):
- Lamar University, Beaumont, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are openly available in Figshare at http://doi.org/10.6084/m9.figshare.13718896
Supporting Information: Study Protocol, SAP
Time Frame: Available now
Access Criteria: Data are openly available
URL: http://doi.org/10.6084/m9.figshare.13718896

REFERENCES:
- See also: Study website — http://www.tacklingtinnitus.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 participants screened at baseline and completed informed consent 3 participants were excluded as they did not meet inclusion criteria 11 participants decided not to participate
Period: Overall Study
Arm/Group | Internet-based Cognitive Behavior Therapy
Started | 32
Completed | 22
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 26
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 17
  Ukraine | 2
  Puerto Rico | 2
  Germany | 1
  France | 1
  Brazil | 6
  Mexico | 2
  Costa Rica | 1
Tinnitus Functional Index (TFI); Measure of Tinnitus Distress [Mean (Standard Deviation); unit: score on a scale] | 61.06 (19.03)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index (TFI); Measure of Tinnitus Distress
Description: Tinnitus Functional Index (TFI) is a 25-item questionnaire that evaluates the severity of tinnitus distress. Total possible score ranges from 0-to-100 with higher scores suggesting more severe tinnitus distress (i.e., worse outcome). Scores >25 indicate tinnitus is a significant problem requiring tinnitus intervention.
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: 32 participants started the trial 22 participants completed the post-intervention measures 16 participants completed the 2-month post-intervention measures
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  Baseline | 61.06 (19.03)
  Post-intervention: number analyzed (Participants) | 22
  Post-intervention | 41.78 (27.02)
  2-months post-intervention: number analyzed (Participants) | 16
  2-months post-intervention | 40.38 (26.65)

2. Secondary Outcome: Tinnitus Cognition Questionnaire (TCQ); Measure of Tinnitus Cognition
Description: Tinnitus Cognition Questionnaire (TCQ) is a 26-item questionnaire that assesses positive and negative cognitions associated with tinnitus. The first 13 items refer to negative thoughts and the second 13 items refer to positive thoughts. Responses are marked on a five-point Likert scale (0 to 4). The negative items (1-13) are scored 0-4, whereas the positive items (14-26) are reverse-scored: 4-0. The scoring procedure involves the simple addition of the number circled by the respondent for items 1-13 and the addition of reverse-scored items 14-26. The total score of the TCQ has a potential range from 0 to 104. A high score represents a greater tendency to engage in negative cognitions (i.e., worse outcome) in response to tinnitus and low engagement in positive cognitions.
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 52.56 (13.18)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 38.55 (24.57)
  T2: 2-month post-intervention: number analyzed (Participants) | 16
  T2: 2-month post-intervention | 37.06 (23.53)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-9); Measure of Depression
Description: Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that assesses depression severity. Responses are marked on a four-point Likert scale (0 to 3). The total score can range from 0 to 27 with higher scores indicating more severe depression (i.e., worse outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 11.25 (7.02)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 5.41 (5.82)
  T2: 2-month post-intervention: number analyzed (Participants) | 16
  T2: 2-month post-intervention | 6.13 (8.55)

4. Secondary Outcome: Generalized Anxiety Disorder (GAD-7); Measure of Anxiety
Description: Generalized Anxiety Disorder (GAD-7) is a 7-item questionnaire that assesses the severity of anxiety. Responses are marked on a four-point Likert scale (0 to 3). The total score can range from 0 to 21 with higher scores indicating more severe anxiety (i.e., worse outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 10.25 (5.32)
  T1: Post-intervention | 5.23 (4.24)
  T2: 2-month post-intervention | 5.62 (5.4)

5. Secondary Outcome: Insomnia Severity Index (ISI); Measure of Insomnia
Description: Insomnia Severity Index (ISI) is a 7-item questionnaire that evaluates insomnia. Responses are marked on a five-point Likert scale (0 to 4). The total score can range from 0 to 28 with higher scores indicating more severe insomnia (i.w., worse outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 14.97 (6.6)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 10.55 (7.11)
  T2: 2-month post-intervention: number analyzed (Participants) | 16
  T2: 2-month post-intervention | 9.38 (7.71)

6. Secondary Outcome: EuroQol EQ-5D-5L VAS; Measure of Health-related Quality of Life
Description: EQ-5D-5L VAS is a single-item questionnaire that evaluates the health-related quality of life. Responses are marked on a 0-100 scale with higher scores indicating higher health-related quality o life (i.e., better outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 67.03 (16.94)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 73.64 (14.65)
  T2: 2-month post-intervention: number analyzed (Participants) | 16
  T2: 2-month post-intervention | 76.75 (15.33)

7. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Tinnitus Sub-scale; Measure of Tinnitus Problem
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problem and ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 16 with higher scores indicating more tinnitus problem (i.e., worse outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 8.06 (3.6)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 4.64 (3.75)
  T2: 2-months post-intervention: number analyzed (Participants) | 16
  T2: 2-months post-intervention | 4.44 (4.35)

8. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Hearing Sub-scale; Measure of Hearing Problem
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problem and ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 16 with higher scores indicating more hearing problem (i.e., worse outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 5.34 (4.29)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 5.55 (4.06)
  T2: 2-months post-intervention: number analyzed (Participants) | 16
  T2: 2-months post-intervention | 3.94 (4.40)

9. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Sound Tolerance Sub-scale; Measure of Sound Tolerance
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problem and ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 8 with higher scores indicating more sound tolerance problem (i.e., worse outcome).
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet-based Cognitive Behavior Therapy
Number analyzed (Participants) | 32
score on a scale
  T0: Baseline | 1.72 (1.28)
  T1: Post-intervention: number analyzed (Participants) | 22
  T1: Post-intervention | 1.5 (1.47)
  T2: 2-months post-intervention: number analyzed (Participants) | 16
  T2: 2-months post-intervention | 1.13 (1.09)

ADVERSE EVENTS:
Time Frame: T0: Baseline, T1: Post-intervention (8-weeks from baseline), T2: 2-months post-intervention (16-weeks from baseline)
Description: Our definition of adverse events is the same as clinical trials.gov.
Arm/Group | Internet-based Cognitive Behavior Therapy
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
The study was done during the height of the COVID-19 pandemic, during a time where day-to-day living was disrupted for most people. This may have been one of the key reasons for poor engagement with the intervention and poor compliance with the completion of outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT04335929/Prot_SAP_000.pdf